CLINICAL TRIAL: NCT02535598
Title: Therapy Labs: To Improve Adherence in Internet Based Psychotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single
Other Study IDs: sveal1031
Record Dates: First submitted 2015-08-03; First posted 2015-08-28 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Behavior Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Normal presentation (Active Comparator): Standard internet based CBT presentation.
  Interventions: Behavioral: Normal presentation
- Enhanced presentation (Experimental): Enhanced internet CBT presentation.
  Interventions: Behavioral: Enhanced presentation
- Normal support (Active Comparator): Standard internet based CBT support.
  Interventions: Behavioral: Normal support
- Enhanced support (Experimental): Enhanced internet CBT support.
  Interventions: Behavioral: Enhanced support

INTERVENTIONS:
Behavioral: Normal presentation — All the material will be presented as plain text.
  Arms: Normal presentation
Behavioral: Enhanced presentation — The material of the intervention is designed to be as appealing as possible with clear organization, animated presentations, ample illustrations, etc.
  Arms: Enhanced presentation
Behavioral: Normal support — Participants receive semi-standardized support once a week and there will be no formal training or competence.
  Arms: Normal support
Behavioral: Enhanced support — Participants are offered daily support through the internet from trained therapists.
  Arms: Enhanced support

SUMMARY:
This project aims to investigate factors that are important in affecting adherence in internet based Cognitive Behavior Therapy (CBT). It is hypothesized that two intervention-specific variables, Support and Content, are important factors and that maximizing the impact of these would result in improved adherence and potentially in the end also better outcome for participants in internet interventions.

DETAILED DESCRIPTION:
This study centers on people with mild symptoms of stress or worry. Participants are recruited by advertisement and the web. Potential participants are contacted by phone and informed about the study. Written informed consent is collected through mail from those who are interested in participating. They are asked to answer all the instruments of the study via a secure internet portal used for delivering the intervention. If they do not fulfill the exclusion criteria they are randomized to one of four conditions. When the intervention has ended participants are asked to fill out all the instruments and again at four week follow up. To find significant (p<.05) results on the primary outcome variables with estimated medium effect sizes, pair-wise comparisons, a power of .80 and allowing for 10% attrition, forty participants are needed in each condition.

The intervention used in this project will be a standard program of applied relaxation that has been used and empirically tested in previous clinical studies. Since the aim of the present project is to investigate factors that affect adherence rather than the intervention effect, the investigators will use a well tested intervention with known effects on symptoms of stress and anxiety. Previous studies have shown that self help with applied relaxation can have a positive effect on for example stress, anxiety and sleep. By providing an intervention that is beneficial, credible and relevant for people with mild symptoms of stress and anxiety it would be possible to investigate how manipulating different factors of the intervention affects the adherence. Applied relaxation will in this intervention consist of a four-week program provided via the Internet. The exact composition of the intervention will be slightly different in each condition depending on the research question, see below. The program includes four steps; tension sensitivity training, long relaxation, short relaxation and applied relaxation. Each week includes information, assignments and support via the secure internet portal.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported mild to moderate symptoms of stress or worry

Exclusion Criteria:

* insufficient mastery of Swedish language
* elevated symptoms of anxiety or depression that warrant clinical care
* other medical or mental illness that need immediate clinical attention
* no daily access to computer, internet and cell phone

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2014-05; Primary Completion 2015-01 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Number of treatment components completed | Four weeks after treatment start
Number of behavioral prescriptions completed | Four weeks after treatment start

SECONDARY OUTCOMES:
Perceived Stress Scale | Baseline and four weeks after treatment start

OTHER OUTCOMES:
Perceived Stress Scale | Baseline and eight weeks after treatment start

CONTACTS AND LOCATIONS:
Overall Officials: Timo Hursti, PhD, Study Director — Uppsala University
Locations (1):
- Uppsala University, Uppsala, Uppsala County, Sweden

REFERENCES:
- [Derived] Alfonsson S, Olsson E, Hursti T. Motivation and Treatment Credibility Predicts Dropout, Treatment Adherence, and Clinical Outcomes in an Internet-Based Cognitive Behavioral Relaxation Program: A Randomized Controlled Trial. J Med Internet Res. 2016 Mar 8;18(3):e52. doi: 10.2196/jmir.5352. PMID 26957354